CLINICAL TRIAL: NCT04633057
Title: A Phase III, Randomized, Open-label, Positive-controlled, Multi-center Study to Evaluating the Efficacy and Safety of Recombinant Long-acting Human Growth Hormone (TJ101) in Children With Growth Hormone Deficiency
Brief Title: A Study to Evaluating the Efficacy and Safety of Recombinant Long-acting Human Growth Hormone (TJ101) in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTJ101PGHD301
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Growth Hormone Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJ101 (Experimental): TJ101 1.2 mg/kg once a week for 52weeks
  Interventions: Drug: TJ101
- NordiFlex (Active Comparator): NordiFlex Injection 0.034 mg/kg once a day for 52 weeks
  Interventions: Drug: NordiFlex

INTERVENTIONS:
Drug: TJ101 — TJ101/ Recombinant Human Somatropin Injection treatment: after screening, subjects will be randomized to receive TJ101 1.2 mg/kg once a week until 52 weeks back site, investigator evaluate effectiveness and safety.
  Arms: TJ101
Drug: NordiFlex — TJ101/ Recombinant Human Somatropin Injection treatment: after screening, subjects will be randomized to receive Recombinant Human Somatropin Injection 0.034 mg/kg once a day, until 52 weeks back site, investigator evaluate effectiveness and safety.
  Arms: NordiFlex

SUMMARY:
A Phase III, Randomized, open-label, positive-drug parallel control, Study to Evaluate the Efficacy and Safety of TJ101 in Child subject with growth hormone deficieney.

ELIGIBILITY:
Inclusion Criteria:

1. Boys: 3 years ≤ boy's age ≤ 10 years；Girls: 3 years ≤ girl's age ≤ 9 years
2. Pre-pubertal children(Tanner stage I)
3. GHD confirmed by 2 different GH provocation tests with peak GH concentration below 10 ng/mL in screening or one month
4. Height (HT) of at least 2.0 standard deviations (SD) below the mean height for chronological age (CA) and gender according to Table of standard deviation unit values of age and height of Chinese children aged 3-12 years , (HT SDS ≤ -2.0)
5. Height velocity≤5.0cm/years (Including height records before at least three months)；
6. IGF-1 SDS≤-1.0
7. Bone age (BA) is no more than two chronological age
8. Body mass Index (BMI) must be within ±2 SD of mean BMI for the chronological age and sex according to Table of standard deviation unit values of Age and BMI of Chinese children aged 3-12 years
9. Without prior exposure to any rhGH therapy
10. For children with growth hormone deficiency that is one of its multiple pituitary hormone deficiencies, alternative therapies targeting the hypothalamus-pituitary-target gland axis must be used for at least 3 months before screening
11. Written informed consent of the parent or legal guardian of the subject and assent of the subject (if the subject can read)

Exclusion Criteria:

1. beyond physiological dosage of glucocorticoid therapy
2. Evidence of closed epiphyses
3. Any other chronic condition that can cause short stature and cannot be treated with hormone replacement therapy(Including but not limited Chronic kidney disease, malnutrition, absorption disorders, uncontrolled hypothyroidism, celiac disease, rickets and social-psychological dwarfism)
4. Abnormal liver and renal function (ALT>1.5 times the upper limit of normal range and Cr exceeding the upper limit of normal range)
5. Presence of anti-hGH antibodies at screening
6. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids, with the exception of ADHD(attention deficit hyperactivity disorder) drug hormone replacement therapies [thyroxine, hydrocortisone, desmopressin (DDAVP)]
7. Mutations in growth hormone receptors are suspected, or any syndrome that causes insensitivity to growth hormone
8. At screening, ophthalmologic examination (including fundus microscopy) indicated increased intracranial pressure and/or retinopathy.
9. At screening, previous or existing intracranial tumor growth was confirmed by cranial magnetic resonance imaging (MRI) scan (using contrast agent) (MRI results up to 1 year prior to screening were acceptable)
10. Diseases such as severe cardiopulmonary, blood system, malignant tumor or potential tumor (family history), or systemic infection, low immune function and mental diseases
11. Significant spinal abnormalities, including scoliosis (Cobb Angle & GT;60 ˚), kyphosis and spina bifida.
12. Subjects diagnosed with type 2 or type 1 diabetes who were considered to have received no standard treatment, did not follow their prescribed treatment, or exhibited poor metabolic control, or had fasting glucose > 5.6 mmol/L twice in a row
13. Chromosomal abnormalities and medical syndromes (Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, SHOX mutations/deletions and skeletal dysplasias), with the exception of septo-optic dysplasia
14. Children with low birth weight (birth weight and/or body length are 2 SD below average according to the standard of the general Chinese population of the same gestational age and sex)
15. The subject and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct
16. Subject who has received an investigational product or has participated in a clinical study within 30 days before screening or during the clinical trials.
17. Known or suspected to be HIV positive, serologically positive for syphilis, or other chronic infectious diseases, such as AIDS, tuberculosis, hepatitis, etc
18. The history of drug, drug or alcohol abuse
19. Other conditions not considered suitable for inclusion by the researchers

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The Annualized Height velocity at 52 week | 52weeks after first dose
  The Annualized Height velocity at 52 week

SECONDARY OUTCOMES:
change in Annualized Height velocity at 26 week (compared to Baseline value) | 26weeks after first dose
change in Annualized Height velocity at 52 week (compared to Baseline value) | 52weeks after first dose

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital, Capital Institute of Paediatrics, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Wanzhou, Chongqing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yet-sen University, Guangzhou, Guangdong
  - Liuzhou Maternity and Children Healthcare Hospital, Liuchow, Guangxi
  - Hainan Third People's Hospital, Sanya, Hainan
  - Tangshan Women and Children's Hospital, Tangshan, Hebei
  - Henan Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jiangsu Provincial Maternal and Child Health Hospital, Nanjing, Jiangsu
  - Children's Hospital affiliated to Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Pingxiang Maternity and Child Care Hospital, Pingxiang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Linyi Women and Children's Hospital, Linyi, Shandong
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Taizhou First People's Hospital, Liuzhou, Zhejiang
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang